CLINICAL TRIAL: NCT01765465
Title: Effect of Rowachol on Prevention of Postcholecystectomy Syndrome After Laparoscopic Cholecystectomy
Brief Title: Effect of Rowachol on Prevention of Postcholecystectomy Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DongGuk University (Other)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, In Woong Han, Assistant Professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-2012-E0816-00001
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Postcholecystectomy Syndrome
Keywords: postcholecystectomy syndrome; laparoscopic cholecystectomy; Rowachol
MeSH Terms: conditions — Postcholecystectomy Syndrome | interventions — Rowachol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rowachol (Experimental): Rowachol treatment with 200mg PO tid, on postoperative 1 days to 3 months
  Interventions: Drug: Rowachol
- Placebo (Placebo Comparator): Placebo treatment with 200mg PO tid, on postoperative 1 days to 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rowachol
  Arms: Rowachol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Postcholecystectomy syndrome (PCS) includes a heterogeneous group of diseases, usually manifested by the presence of abdominal symptoms following gallbladder removal. The pathogenesis of PCS has not been identified; therefore there is no consensus of medical treatment on PCS. The Action of Rowachol are to inhibit hepatic 3-hydroxy-3-methylglutaric acid(HMG)-coenzyme A(CoA) reductase, to inhibits cholesterol nucleation in bile from patients with cholesterol gallstones, and to promote biliary lipid secretion.

The purpose of this study is to determine whether Rowachol is useful in the prevention of PCS and symptoms change after laparoscopic cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologic diseases scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Current immunosuppressive therapy
* Chemotherapy within 4 weeks before operation
* Radiotherapy completed longer than 4 weeks before operation
* Inability to follow the instructions given by the investigator
* Severe psychiatric or neurologic diseases
* Drug- and/or alcohol-abuse according to local standards
* Participation in another intervention-trial with interference of a primary or secondary endpoint of this study
* Lack of compliance
* Lack of informed consent

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In Woong Han, M.D., Principal Investigator — DongGuk University College of Medicine
Locations (2):
- South Korea (2):
  - DongGuk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Chung-Ang University Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Rowachol: Rowachol treatment with 200mg PO tid, on postoperative 1 days to 3 months
  Rowachol
- Placebo: Placebo treatment with 200mg PO tid, on postoperative 1 days to 3 months
  Placebo
Period: Overall Study
Arm/Group | Rowachol | Placebo
Started | 71 | 67
Completed | 64 | 63
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rowachol | Placebo | Total
Number analyzed (Participants) | 71 | 67 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.48 (15.56) | 47.99 (13.81) | 49.78 (14.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 34 | 79
  Male | 26 | 33 | 59

OUTCOME MEASURES:

1. Primary Outcome: the Number of the Participants Have Postoperative RUQ Pain
Description: Right upper quadrant(RUQ) pain by European Organization for Research and Treatment of Cancer(EORTC) quality of life questionnaire(QLQ) C-30 No. 9, 19 at baseline and postoperative 3-month.
  The pain score of individuals at postoperative 3-month is calculated by EORTC QLQ C-30 manual.
  The pain score range is 0 to 100. Higher score means participants feel more pain(worse). If a participant's pain score is over 30, we define he/she has post operative RUQ pain. we use the number of the participants have post operative RUQ pain(score over 30) as the results.
Time Frame: postoperative 3-month
Measure: Number; unit: number of participants
Arm/Group | Rowachol | Placebo
Number analyzed (Participants) | 64 | 63
number of participants | 3 | 9

2. Secondary Outcome: Laboratory Test Results of Postoperative 3-month(Total Bilirubin, Direct Bilirubin)
Description: laboratory test results(liver function test such as total bilirubin, direct bilirubin) measured at postoperative 3-month of Rowachol group and placebo group.
  each result is mean values.
Time Frame: postoperative 3-month
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Rowachol: Rowachol treatment with 200mg PO tid, on postoperative 1-day to 3-month
  Rowachol
- Placebo: Placebo treatment with 200mg PO tid, on postoperative 1-day to 3-month
  Placebo
Arm/Group | Rowachol | Placebo
Number analyzed (Participants) | 64 | 63
mg/dL
  Total bilirubin | 0.7 (0.5) | 0.6 (0.2)
  Direct bilirubin | 0.3 (0.3) | 0.2 (0.2)

3. Secondary Outcome: Laboratory Test Results of Postoperative 3-month(Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase)
Description: laboratory test results(liver function test such as Alkaline phosphatase, Aspartate aminotransferase, Alanine aminotransferase) measured at postoperative 3-month of Rowachol group and placebo group.
  each result is mean values.
Time Frame: postoperative 3-month
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Rowachol | Placebo
Number analyzed (Participants) | 64 | 63
IU/dL
  Alkaline phosphatase | 242.8 (449.8) | 209.6 (145.5)
  Aspartate aminotransferase | 105.1 (60.5) | 50.8 (41.2)
  Alanine aminotransferase | 44.3 (43.8) | 56.1 (49.1)

4. Secondary Outcome: Laboratory Test Results of Postoperative 3-month(WBC Count)
Description: laboratory test results(WBC count) measured at postoperative 3-month of Rowachol group and placebo group.
  each result is mean values.
Time Frame: postoperative 3-month
Measure: Mean (Standard Deviation); unit: cells (10^6/µl)
Arm/Group | Rowachol | Placebo
Number analyzed (Participants) | 64 | 63
cells (10^6/µl) | 6.8 (2.1) | 7.2 (2.4)

ADVERSE EVENTS:
Time Frame: postoperative 3 months
Arm/Group | Rowachol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 1/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rowachol (N=64) | Placebo (N=63)
Post operative minor bile leak (Hepatobiliary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No